CLINICAL TRIAL: NCT04968938
Title: A Phase 2, Open Label Study of the Safety and Effectiveness of MDMA-assisted Therapy for Participants With Posttraumatic Stress Disorder
Brief Title: Study of Safety and Effects of MDMA-assisted Therapy for Treatment of PTSD
Acronym: NUMCAP1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decided not to pursue the study. Study ended prior to study start.
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NUMCAP1
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MDMA-assisted therapy (Experimental): Two sessions of MDMA-assisted therapy with an initial dose of 80 mg or 120 mg midomafetamine HCl and optional supplemental dose of 40 mg 1.5 to 2 hours later
  Interventions: Drug: midomafetamine; Behavioral: Therapy

INTERVENTIONS:
Drug: midomafetamine — 80 mg or 120 mg midomafetamine HCl followed by a 40 mg supplement dose
  Other Names: MDMA; midomafetamine HCl
Behavioral: Therapy — Manualized therapy

SUMMARY:
The purpose of this clinical trial is to learn if MDMA-assisted therapy is safe and effective in people with PTSD.

The main question it aims to answer is: Do two open-label sessions of MDMA-assisted therapy reduce PTSD symptoms?

Participants will undergo three non-drug preparatory therapy sessions followed by two open-label MDMA-assisted therapy sessions. After, participants will undergo three non-drug integrative therapy sessions.

DETAILED DESCRIPTION:
This Phase 2, open-label study will provide supportive data on the safety and effectiveness of MDMA-assisted therapy in participants with PTSD. This study will be conducted at a single study site in Vancouver, BC. There will be at least 2 co-therapy pairs. The study will enroll up to 20 participants.

The Preparatory Period will consist of three 90-minute non-drug preparatory therapy sessions. A flexible divided dose of MDMA will be administered during the Treatment Period with manualized therapy in up to two open-label experimental sessions. During the Treatment Period, each experimental session is followed by three 90-minute non-drug integrative therapy sessions. The experimental sessions are scheduled roughly 3 to 5 weeks apart.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years old.
* Are fluent in speaking and reading a recognized language of the study site.
* Are able to swallow pills.
* Agree to have study visits recorded, including Study Drug Sessions and non-drug therapy sessions.
* Must provide a contact (relative, spouse, close friend, or other support person) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable.
* Must agree to inform the investigators within 48 hours of any medical conditions and procedures.
* If of childbearing potential, must have a negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate birth control through 10 days after the last Experimental Session.
* Must not participate in any other interventional clinical trials during the duration of the study, and commit to medication dosing, therapy, and study procedures.
* At baseline, have moderate PTSD diagnosis.

Exclusion Criteria:

* Are not able to give adequate informed consent.
* Have uncontrolled hypertension.
* Have a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds [ms] in males and>460 ms in females corrected by Friderica's formula).
* Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
* Have evidence or history of significant medical disorders.
* Have symptomatic liver disease.
* Have history of hyponatremia or hyperthermia.
* Weigh less than 48 kilograms (kg).
* Are pregnant or nursing, or are of childbearing potential and are not practicing an effective means of birth control.
* Have current alcohol or substance use disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in PTSD Checklist (adapted PCL-5) total score | 18 weeks post baseline post enrollment confirmation
  20-item self-report questionnaire in which respondents indicate the presence and severity of PTSD symptoms, derived from the symptoms of PTSD per DSM-5. The gold standard for diagnosing PTSD is a structured clinical interview such as the Clinician-Administered PTSD Scale (CAPS-5). When necessary, the PCL-5 can be scored to provide a provisional PTSD diagnosis.The self-report rating scale is 0-4 for each symptom, reflecting a change from 1-5 in the DSM-IV version. Rating scale descriptors are the same: "Not at all," "A little bit," Moderately," "Quite a bit," and "Extremely."

CONTACTS AND LOCATIONS:
Overall Officials: Devon Christie, MD, Principal Investigator — Department of Medicine, University of British Columbia

IPD SHARING:
Plan to Share IPD: Yes
We will share outcome data appearing in any published reports upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data and study-related documents will be available when the database has been locked and data has been unblinded.
Access Criteria: Interested persons should correspond with the central contact for the multisite study.